CLINICAL TRIAL: NCT00374426
Title: Preventing Depression Recurrence in Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96-0806 (completed); DK53060
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Major Depression; Diabetes
Keywords: depression; diabetes mellitus; depression recurrence
MeSH Terms: conditions — Depressive Disorder, Major; Diabetes Mellitus; Depression | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline

SUMMARY:
To study the effectiveness of sertraline (Zoloft) in treating depression in adults with diabetes. The study will also determine whether depressed diabetic patients who have successfully responded to sertraline (Zoloft) are more likely to have depression recur if the sertraline (Zoloft) is discontinued.

DETAILED DESCRIPTION:
Part A: Prevention of Depression Recurrence in Diabetes

1. To determine the efficacy of maintenance antidepressant medication in preventing or delaying recur-rence of major depression in diabetes.
2. To determine the relationship of sustained depression remission to social, occupational, and global func-tioning, and to quality of life and compliance with diabetes treatment.
3. To determine clinical features predictive of depression recurrence in diabetes.

Part B. Longitudinal Study of the Interrelationship of Glycemic Control and Depression

1. To determine the effects of depression remission and recurrence on glycemic control.
2. To determine the efficacy of maintenance antidepressant medication in producing sustained benefits in glycemic control.
3. To determine the interrelationship of daily mood with blood glucose and the effect of maintenance treatment on this relationship.

ELIGIBILITY:
Inclusion Criteria:

* 18-80
* Type 1 or Type 2 Diabetes
* Screen positive for depression

Exclusion Criteria:

* Are pregnant or lactating
* Are known to be hypersensitive to the drug
* Have a recent history of myocardial infarction or unstable heart disease
* Have severe hepatic disease or renal impairment (serum creatinine > 3 mg/dl)
* The subset of patients with psychiatric disorders thought to affect management (e.g., schizophrenia, alcohol and drug dependence) will also be excluded from participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262
Dates: Start 1998-03; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Lustman, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States